CLINICAL TRIAL: NCT02264873
Title: Minimizing Leukemia Relapse: A Phase I, Dose Escalation Study of Decitabine in High Risk Pediatric Leukemia Post Allogeneic Transplant
Brief Title: Phase I, Dose Escalation Study of Decitabine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Hyundai Hope On Wheels (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201400612; PEDS004 (Other: University of Florida Protocol ID)
Record Dates: First submitted 2014-10-06; First posted 2014-10-15 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Leukemia, Lymphoblastic, Acute; Leukemia, Myeloid Acute; Hematopoetic Myelodysplasia
Keywords: Relapse; Autologous stem cell transplant
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Recurrence | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine (Other): This is a 3+3 design of dose escalation
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Dose escalation starting at 5 mg, and increasing by 2.5 mg to a Dose Level of 12.5 mg qd x 3 days.
  Other Names: Decitabine, Dacogen

SUMMARY:
Decitabine is a hypomethylating agent that has shown significant anti-leukemic effect in Myelodysplastic Syndrome (MDS) and Acute Myeloblastic Leukemia (AML). This study is based on the hypothesis that Decitabine delivered after allo-hematopoietic stem cell transplant (HSCT) in patients with leukemia will enhance disease control by the allogeneic immune system and lead to a longer disease free survival. The study is designed to provide safety data of low-dosing in the post-transplant setting.

DETAILED DESCRIPTION:
Decitabine is a hypomethylating agent with significant anti-leukemic effect in MDS and AML. Additionally, aberrant DNA methylation has been identified in high risk childhood ALL, and therefore, DNA hypomethylating agents, such as decitabine, have been identified as therapeutic agents. Moreover, decitabine has immunomodulatory effects by enhancement of class I human leukocyte antigen (HLA) antigen expression on cancer cells, which increases their susceptibility to immune surveillance mechanisms, such as graft-versus-leukemia effect of donor cells in allogeneic transplantation and by augmentation of natural killer (NK), T and B lymphocyte reactivity. We hypothesize that decitabine delivered after allo-HSCT in patients with leukemia will enhance disease control by the allogeneic immune system and lead to a longer disease free survival. However, a safety study is needed to determine appropriate decitabine dosing in the post-transplant period. Low doses of decitabine are likely better tolerated in the post-transplant setting given risks of myelosuppression. In addition, when administered at lower doses, decitabine's hypomethylation effects are more pronounced in relation to its pyrimidine analog cytotoxic effects. In this study low doses of decitabine will be administered beginning 6 weeks to 100 days post-transplant. Measures of gene methylation and immune reconstitution will be conducted to define biologically active doses. Results from this trial will provide new clinical data regarding the effects of decitabine on gene methylation and immunoreactivity, will establish a maximally tolerated dose in the post-transplant setting, will define biologically active doses, and will serve as a basis for future efficacy trials.

ELIGIBILITY:
Inclusion Criteria:

* Age: greater than 1 and less than 31 years of age;
* Diagnosis: history of ALL, AML or MDS, currently in a complete remission (CR) following allo-HSCT (bone marrow leukemic blasts less than 5% by morphology), with high risk features including:
* Status post allogeneic HSCT
* GVHD prophylaxis:
* Karnofsky or Lansky performance scores more than 50%. Karnofsky scores will be used for patients > 16 years of age and Lansky scores for patients ≤ 16 years of age;
* Platelet count ≥ 50,000 (untransfused);
* Absolute neutrophil count ≥ 1000; and;
* Hemoglobin ≥ 8 g/dL (un-transfused);

Exclusion Criteria:

* Progressive disease;
* Philadelphia chromosome positive ALL (these patients receive tyrosine kinase inhibitor posttransplant);
* Known hypersensitivity to any components of decitabine;
* Uncontrolled grade 3-4 graft versus host disease;
* Uncontrolled infection;
* Serum creatinine > 2 mg/dL or glomerular filtration rate (GFR) less than 60 mL/min/1.73m2 ;
* Alanine Aminotransferase (ALT) greater than 3 times normal or serum total bilirubin greater than 2 mg/dL;

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose as a Measure of Safety and Tolerability | 3 months
  This is a dose escalation study of decitabine maintenance therapy after allo-HSCT for the maximally tolerated dose in pediatric patients without adverse events.

SECONDARY OUTCOMES:
Adverse Event Profile After Single Cycle Decitabine Post Transplant | 6 months
  The adverse events will be graded using the NCI Scale after one cycle of decitabine maintenance therapy intravenously. Grade 1 and 2 are unexpected and expect but unlikely related or unrelated; Grade 3 unexpected with hospitalization within 10 calendar days or possibly, probable related and without hospitalization; Grade 3 expected with hospitalization within 10 days or without hospitalization; Grade 4 and 5 Unexpected and Expected 24-hours to 5 days unlikely, unrelated, possible, probable, definite.
Grade 3 Adverse Events after Decitabine | 6 months
  To estimate the incidences of ≥ grade 3 adverse events, infections, need for transfusions, treatment related mortality (TRM), and incidence and severity of graft vs host disease (GVHD) after initiation of decitabine post-HSCT. The grading will be done with the NCI Scale Grade 3 unexpected with hospitalization within 10 calendar days or possibly, probable related and without hospitalization; Grade 3 expected with hospitalization within 10 days or without hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Castillo, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Hospital, Gainesville, Florida, United States